CLINICAL TRIAL: NCT00679224
Title: A Post-Marketing Observational Surveillance Programme for Ambrisentan (VOLT)
Brief Title: An Observational Study For Ambrisentan
Acronym: VOLT
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110094
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertesion; observational safety
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ambrisentan prescribed subjects: ambrisentan prescribed subjects
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — ambrisentan

SUMMARY:
The purpose of the programme is to collect safety data on ambrisentan when used in clinical practice

DETAILED DESCRIPTION:
The purpose of the programme is to collect safety data on ambrisentan when used in clinical practice

ELIGIBILITY:
subjects who have been prescribed ambrisentan for a medically appropriate use (see approved product label)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects who have been prescribed ambrisentan for a medically appropriate use. (See approved product label e.g. Summary of Product Characteristics. )
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
safety monitoring

SECONDARY OUTCOMES:
safety monitoring

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (102):
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Aarhus N, Denmark
- France (20):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (26):
  - GSK Investigational Site, Donaueschingen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Gerlingen, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Löwenstein, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Treuenbrietzen, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (4):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Voula / Athens
- Italy (9):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
- Netherlands (6):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
- Spain (9):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Ourense
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Valencia
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
- United Kingdom (5):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield